CLINICAL TRIAL: NCT02822027
Title: Intravenous Immunoglobin Transfusion in Preterm Infants With Encephalopathy of Prematurity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Fang Wu, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVIG for encephalopathy
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Preterm Infants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- human gamma globulin (Experimental): human gamma globulin for infants with encephalopathy of prematurities
  Interventions: Drug: human gamma globulin; Drug: non-human gamma globulin
- non-human gamma globulin (Active Comparator): non-human gamma globulin for infants with encephalopathy of prematurities
  Interventions: Drug: human gamma globulin; Drug: non-human gamma globulin

INTERVENTIONS:
Drug: human gamma globulin — human gamma globulin for preterm infants with encephalopathy of prematurities
Drug: non-human gamma globulin — Non-human gamma globulin for preterm infants with encephalopathy of prematurities

SUMMARY:
Infection and inflammation is related to increased encephalopathy of prematurities.

DETAILED DESCRIPTION:
Animal studies have verified intravenous immunoglobin can reduce brain injury. However, no studies in preterm infants were reported.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with encephalopathy

Exclusion Criteria:

* refuse the participate in the trial

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
structural changes of brain injury | 100-days
  MRI/ultrasound will be used to assess the structural severities of brain injury.
functional changes of brain injury | 100-days
  Bayley score will be used to assess the functional severities of brain injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics,Daping Hospital, Chongqing, Chongqing Municipality, China